CLINICAL TRIAL: NCT05533515
Title: Circulating Tumour Cells as Biomarkers to Predict Prostate Cancer Metastasis for Treatment Stratification of Localised Cancer
Brief Title: Circulating Tumour Cells as Biomarkers to Predict Prostate Cancer Metastasis for Treatment Stratification of Cancer
Acronym: C-ProMeta-1
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 19/LO/0994; 140998 (Other: IRAS)
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 x 10 ml blood samples will be collected (months 1-27) using the lavender cap EDTA tube according to our established method from each consented patient by the CRF or the clinical care team at UCLH during the pre- and post-RP PSA test blood sampling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RP Treatment cohort: We will use participants who have been deemed eligible for radical prostatectomy based on the current European Urology Association classification system, and who have been scheduled for surgery to completely remove the cancer in the prostate gland.
  Interventions: Diagnostic Test: CTC Blood Test

INTERVENTIONS:
Diagnostic Test: CTC Blood Test — We will draw blood to measure the level of Circulating Tumour Cells

SUMMARY:
The goal of this study is to establish the value of Circulating Tumour Cell (CTC) positivity in predicting post-RP treatment failure, including BCR and new lesions detected by cancer imaging. We plan to recruit participants who will undergo Radical Prostatectomy (RP). Participants will have their blood samples taken just before surgery and 3 months after the surgery to test for CTCs. Then participants will be followed-up for cancer progression information at 3 month intervals for the first year then yearly intervals after that. Their PSA will be observed over time.

DETAILED DESCRIPTION:
This is a single site, double-blinded, prospective, paired cohort study. Participating patients and clinicians involved in treatment or management will be blinded to the CTC results, to avoid influencing standard patient treatment, management, and progression outcomes after RP.

Patients will be recruited (months 1-24) at UCLH, where the UK largest urological surgery centre is located and performs robot-assisted RP on PCa patients referred from several regional hospitals. The clinical team at UCLH will identify eligible patients who will be approached by the clinical research fellow (CRF) employed on the research project or the clinical care team for informed consent using the consent forms specifically designed for this project for blood collection and future research. Non-metastatic disease will be based on the current standard diagnostic imaging methods including CT/MRI and PSMA-PET/bone scan. A pre-surgery PSA test will be performed routinely at UCLH.

2 x 10 ml blood samples will be collected (months 1-27) using the lavender cap EDTA tube according to our established method from each consented patient by the CRF or the clinical care team at UCLH during the pre- and post-RP PSA test blood sampling, and taken to the laboratory at Barts Cancer Institute, John Vane Science Centre, Charterhouse Square either by the CRF, a tissue bank acquisition officer (TBAO)(in the absence of the CRF) or the postdoc (anonymise samples transfer in the absence of CRF and TBAO) under the signed material transfer agreement (MTA), at room temperature. The samples will be transported in designated sample carrier using a taxi service. No public transport is to be used for moving samples between sites.

ELIGIBILITY:
Inclusion Criteria:

* High/High intermediate risk non-metastatic risk localised PCa based on the EAU stratification system
* Scheduled for robot-assisted RP
* Informed consent

Exclusion Criteria:

* With other co-occurring cancers
* Neo-adjuvant ADT
* Adjuvant ADT

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to recruit patients meeting the eligibility criteria, it will be necessary to screen all patients in the participating centre who are diagnosed with high risk localised PCa based on the current European Urology Association classification system and who have been scheduled for surgery to completely remove the cancer in the prostate gland.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Post-RP treatment failure during the first 4.5 years of follow up from start of recruitment. | 4.5 years from the start of recruitment
  Post-RP treatment failure is defined as a PSA ≥ 0.2mg/ml at the routine PSA test 3 months after RP (commonly called 'failure to nadir') and remaining at this level or further increase afterwards without further treatment, or imaging detected appearance of cancer lesions.
  Cancer lesions detected by imaging without a PSA rise might include neuroendocrine PCa and lesions detected by PSAM-PET. This combined post-RP treatment failure primary endpoint will maximally capture all the clinically significant cancer appearance events.

SECONDARY OUTCOMES:
BCR during the first 4.5 years of follow up | 4.5 years
  BCR during the first 4.5 years of follow up: PSA ≥ 0.2ng/ml at any time post-RP and remaining at this level or further increase afterwards without further treatment.
Metastasis free survival (4.5yrs) | 4.5 years
  Metastasis (any location)-free survival during the first 4.5 years of follow up. Only 5% of subjects with distant metastasis event (based on traditional imaging technologies) within this time frame (4-6).
Metastasis free survival (10yrs) | 10 years
  Metastasis (any location)-free survival at 10 years follow up. to confirm that metastatic event rates have increased among the positives, i.e. a declining rate of "false positives".
Deaths (4.5yrs) | 4.5 years
  Deaths from any cause during the first 4.5 years of follow up
10 year survival | 10 years
  Overall survival at 10 years of follow up.
Prostate cancer deaths (4.5yrs) | 4.5 years
  Prostate cancer specific deaths during the first 4.5 years of follow up. Expected to be 2% or less based on previous studies in the post RP context.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Shaw, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We will share the IPD after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as possible after publishing the main study
Access Criteria: Reviewed by study management group for clinical/scientific benefit.

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT05533515/Prot_000.pdf
  • Informed Consent Form (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT05533515/ICF_001.pdf